CLINICAL TRIAL: NCT01031160
Title: Health Behavior in School-Age Children: NEXT Longitudinal Study 2009-2016
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909231; 09-CH-N231
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-09-16

CONDITIONS: Adolescent Health
Keywords: Health Indicators; Health Behaviors; Health Study; Natural History; Substance Abuse; Adolescence; Obesity
MeSH Terms: conditions — Health Behavior; Substance-Related Disorders; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- U.S. high school students: U.S. high school students who were in 10th grade in the 2009-2010 school year.

SUMMARY:
NEXT is a seven-year longitudinal assessment of a representative sample of U.S. adolescent and young adults starting at grade 10. The goals of the NEXT longitudinal study include: to identify the trajectory of adolescent health status and health behaviors from mid-adolescence through the post high school years; to examine individual predictors of the onset of key adolescent risk behaviors and risk indicators during this period; to identify genetic, personal, family, school, and social/environmental factors that promote or sustain positive health behaviors; to identify transition points in health risk and risk behaviors and changes in family, school, and social/environmental precursors to these transitions, and to examine the role of potential gene-environment interactions in the development of health status and health behaviors. .

This study collects reliable and valid data on health behaviors and health indicators and their social, environmental, and biological contexts beginning with a nationally representative probability cohort of 10th-grade children in the U.S in 2009 and following them through 2016. Measures are collected annually for seven years beginning in the 2009-2010 school year and ending in the 2016-2017 school year. African-American youth are oversampled to provide better population estimates of this group and to provide an adequate sample to examine racial/ethnic differences in longitudinal predictors of health, health behaviors, and health behavior change. Hispanic youth do not require oversampling because they currently represent a sufficient proportion of the population of adolescents to provide an adequate sample to examine racial/ethnic differences. Self-reports of health status, health behaviors, and health attitudes are collected by in-school and online surveys. Anthropometric data, genetic information, and neighborhood characteristics are gathered on all participants as well. The study also incorporates an Administrator Survey and other data sources to obtain related information on school-level health programs and community-level contextual data. The NEXT Generation Health Study data support NICHD, National Heart, Lung and Blood Institute (NHLBI), National Institute on Drug Abuse (NIDA), National Institute on Alcohol Abuse and Alcoholism (NIAAA) and the Maternal and Child Health Branch of the Health Resources and Services Administration (HRSA/MCHB) in fulfillment of program requirements that address supportive health environments for adolescents and young adults. In addition, a representative subsample of overweight and normal weight adolescents has been identified: additional data on behavioral risk factors and biological markers and risk factors are gathered on these adolescents. Driving performance will also be evaluated in 150 young adults.

DETAILED DESCRIPTION:
NEXT is a seven-year longitudinal assessment of a representative sample of U.S. adolescent and young adults starting at grade 10. The goals of the NEXT longitudinal study include: to identify the trajectory of adolescent health status and health behaviors from mid-adolescence through the post high school years; to examine individual predictors of the onset of key adolescent risk behaviors and risk indicators during this period; to identify genetic, personal, family, school, and social/environmental factors that promote or sustain positive health behaviors; to identify transition points in health risk and risk behaviors and changes in family, school, and social/environmental precursors to these transitions, and to examine the role of potential gene-environment interactions in the development of health status and health behaviors. .

This study collects reliable and valid data on health behaviors and health indicators and their social, environmental, and biological contexts beginning with a nationally representative probability cohort of 10th-grade children in the U.S in 2009 and following them through 2016. Measures are collected annually for seven years beginning in the 2009-2010 school year and ending in the 2016-2017 school year. African-American youth are oversampled to provide better population estimates of this group and to provide an adequate sample to examine racial/ethnic differences in longitudinal predictors of health, health behaviors, and health behavior change. Hispanic youth do not require oversampling because they currently represent a sufficient proportion of the population of adolescents to provide an adequate sample to examine racial/ethnic differences. Self-reports of health status, health behaviors, and health attitudes are collected by in-school and online surveys. Anthropometric data, genetic information, and neighborhood characteristics are gathered on all participants as well. The study also incorporates an Administrator Survey and other data sources to obtain related information on school-level health programs and community-level contextual data. The NEXT Generation Health Study data support NICHD, National Heart, Lung and Blood Institute (NHLBI), National Institute on Drug Abuse (NIDA), National Institute on Alcohol Abuse and Alcoholism (NIAAA) and the Maternal and Child Health Branch of the Health Resources and Services Administration (HRSA/MCHB) in fulfillment of program requirements that address supportive health environments for adolescents and young adults. In addition, a representative subsample of overweight and normal weight adolescents has been identified: additional data on behavioral risk factors and biological markers and risk factors are gathered on these adolescents. Driving performance will also be evaluated in 150 young adults.

ELIGIBILITY:
* INCLUSION CRITERIA:

Both boys and girls will be recruited for participation in the study. African American youth will be over-sampled to improve population estimates

Study Inclusion Criteria:

All participants previously recruited in the NEXT Generation Health Study are eligible for inclusion in the future assessments.

Next Plus Inclusion Criteria:

Participants are included in the NEXT Plus if they met the criteria for and completed the NEXT survey in Wave 1 and the Wave 1 in-school assessments of height and weight and they and their parents completed the NEXT Plus consent and assent forms.

EXCLUSION CRITERIA:

Survey Exclusion Criteria:

Participants are excluded from participating in the study for any of the following:

* No informed consent from parent(s),
* No informed assent/consent (depending on age) from the participant, or
* Developmental limitations that affect the participant s ability to understand or provide age appropriate responses to the questions posed

Home Visit Exclusion Criteria:

Participants are excluded from participating in NEXT Plus for any of the following:

* No informed consent from parent(s),
* No informed assent/consent from the child,
* Developmental limitations that affect the child s ability to understand or provide age appropriate responses to the questions posed, or
* A blood condition that increases the risk of bleeding.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will include two phases. Phase 1 will include a secondary data analysis with emerging adults and peer driving data acquired from the NEXT Longitudinal Study collected by the National Institute of Child Health and Human Development (NICHD) at the NIH. Phase 2 will include conducting qualitative data collection through 4-5 focus groups on University of Maryland College Park (UMCP) campus with undergraduate students (age 18-22) to understand the influential factors associated with social norms on distracted driving
Sampling Method: Probability Sample
Enrollment: 4902 (Actual)
Dates: Start 2010-02-17 (Actual)

PRIMARY OUTCOMES:
Identify the trajectories of adolescent health and health behaviors, including diet and physical activity, substance use, driving, dating violence, and health status. | baseline
  Identify the trajectories of adolescent health and health behaviors, including diet and physical activity, substance use, driving, dating violence, and health status.

SECONDARY OUTCOMES:
Identify genetic, individual, family, school, social, and other environmental factors that promote or sustain positive health, positive health behaviors and mental health. | ongoing
  Identify genetic, individual, family, school, social, and other environmental factors that promote or sustain positive health, positive health behaviors and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Denise L Haynie, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Protocol does not indicate plans on IPD availability.

REFERENCES:
- [Background] Pratt C, Webber LS, Baggett CD, Ward D, Pate RR, Murray D, Lohman T, Lytle L, Elder JP. Sedentary activity and body composition of middle school girls: the trial of activity for adolescent girls. Res Q Exerc Sport. 2008 Dec;79(4):458-67. doi: 10.1080/02701367.2008.10599512. PMID 19177947
- [Background] HEALTHY Study Group; Hirst K, Baranowski T, DeBar L, Foster GD, Kaufman F, Kennel P, Linder B, Schneider M, Venditti EM, Yin Z. HEALTHY study rationale, design and methods: moderating risk of type 2 diabetes in multi-ethnic middle school students. Int J Obes (Lond). 2009 Aug;33 Suppl 4(Suppl 4):S4-20. doi: 10.1038/ijo.2009.112. PMID 19623188
- [Derived] Yu J, Goldstein RB, Haynie DL, Luk JW, Fairman BJ, Patel RA, Vidal-Ribas P, Maultsby K, Gudal M, Gilman SE. Resilience Factors in the Association Between Depressive Symptoms and Suicidality. J Adolesc Health. 2021 Aug;69(2):280-287. doi: 10.1016/j.jadohealth.2020.12.004. Epub 2021 Jan 9. PMID 33431248
- [Derived] Luk JW, Sita KR, Lewin D, Simons-Morton BG, Haynie DL. Sexual Orientation and Sleep Behaviors in a National Sample of Adolescents Followed Into Young Adulthood. J Clin Sleep Med. 2019 Nov 15;15(11):1635-1643. doi: 10.5664/jcsm.8030. PMID 31739854
- [Derived] Haynie DL, Lewin D, Luk JW, Lipsky LM, O'Brien F, Iannotti RJ, Liu D, Simons-Morton BG. Beyond Sleep Duration: Bidirectional Associations Among Chronotype, Social Jetlag, and Drinking Behaviors in a Longitudinal Sample of US High School Students. Sleep. 2018 Feb 1;41(2):zsx202. doi: 10.1093/sleep/zsx202. PMID 29237053
- [Derived] Lipsky LM, Nansel TR, Haynie DL, Liu D, Li K, Pratt CA, Iannotti RJ, Dempster KW, Simons-Morton B. Diet quality of US adolescents during the transition to adulthood: changes and predictors. Am J Clin Nutr. 2017 Jun;105(6):1424-1432. doi: 10.3945/ajcn.116.150029. Epub 2017 Apr 26. PMID 28446498